CLINICAL TRIAL: NCT03769792
Title: Evaluation of the Effectiveness and Safety of Impedance Spectroscopy Device in Detecting Sphincter Injuries in Women After Natural Delivery
Brief Title: Impedance Spectroscopy in Detection of Obstetric Anal Sphincter Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OASIS Diagnostics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1/1/2018 (Sep 8)
Record Dates: First submitted 2018-10-09; First posted 2018-12-10 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Obstetric Anal Sphincter Injury; Delivery, Obstetric
Keywords: Obstetrical anal sphincter injury; Impedance spectroscopy
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Impedance spectroscopy (Experimental): 24 women will be included in the study and divided into two subgroups.
  12 of them (first subgroup) came from patients within 6 to 8 weeks after natural delivery, that had a perianal tear of grade 1 or 2 in OASIS classification.
  Remaining 12 (second subgroup) came from patients within 6 to 8 weeks after natural delivery, that had a perianal tear of grade 3 or 4 in OASIS classification.
  The planned interventions are:
  * Blood and faeces tests
  * Impedance spectroscopy test
  * Full gynecological and proctological examination
  * Transanal ultrasonography
  * Anorectal manometry
  Interventions: Diagnostic Test: Blood and faeces tests; Device: Impedance spectroscopy test; Diagnostic Test: Full gynecological and proctological examination; Diagnostic Test: Transanal ultrasonography; Diagnostic Test: Anorectal manometry

INTERVENTIONS:
Diagnostic Test: Blood and faeces tests — During V0 - Laboratory tests, particularly for calprotectin concentration assessment
Device: Impedance spectroscopy test — During V1 - the electrical impedance of pelvic floor muscles will be measured
Diagnostic Test: Full gynecological and proctological examination — During V1 - Examination with a gynecological speculum, Two-handed examination, Rectal examination and Anoscopy
Diagnostic Test: Transanal ultrasonography — During V2 - reference diagnostic methods with documented effectiveness and safety; for comparison with impedance spectroscopy results.
Diagnostic Test: Anorectal manometry — During V2 - reference diagnostic methods with documented effectiveness and safety; for comparison with impedance spectroscopy results.

SUMMARY:
The main purpose of the study is to evaluate the effectiveness and safety of the impedance spectroscopy device prototype in detection of anal sphincter injuries in women in the early postpartum period. The study is prospective. The study group comprises 24 patients; included in it 6-8 weeks after natural delivery. The planned participation of each patient in the study is up to 4 weeks and three visits will take place at that time.

After obtaining written consent, at the screening visit (V0) each patient will undergo a physical examination, blood samples for laboratory tests and stool samples for calprotectin concentration assessment will be collected.

On the second visit (V1), after the final verification of inclusion/exclusion criteria, impedance spectroscopy using tested device will be performed in each patient, the electrical impedance of pelvic floor muscles will be measured and the degree of anal sphincter damage will be evaluated. Full gynecological and proctological examination (including a gynecological speculum, two-handed examination, rectal examination and anoscopy) will be carried out.

On the third visit (V2), two reference diagnostic tests (with evidenced effectiveness and safety), transanal ultrasonography and anorectal manometry, will be conducted. The collected data will be used to select the optimal therapeutic method for each participant individually.

ELIGIBILITY:
Inclusion Criteria:

* after natural delivery and post-partum period (6-8 weeks after delivery)
* physiological pregnancy
* observed a perianal tear of grade 1-4 in the OASIS classification
* signed informed consent

Exclusion Criteria:

* presence of acute diseases during treatment
* presence of chronic diseases untreated or insufficiently treated (e.g. poorly controlled hypertension),
* presence of diseases, with symptoms of fecal incontinence,
* previous proctological operations,
* the presence of inflammatory bowel diseases in the stage of exacerbation,
* treatment in the last year due to severe, progressive, uncontrolled cardiac, pulmonary, nephrological, infectious or psychiatric disease, which course could affect the patient's risk due to participation in study,
* significant deviations from the norm in a physical examination during V0 visit or laboratory tests taken during the same visit,
* significant disease symptoms so far undiagnosed and reported during the V0 visit
* presence or suspected malignant disease or previous oncological treatment during the last 5 years,
* presence of a cardiac stimulator or cardioverter-defibrillator,
* severe surgery or severe trauma in the last year.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Anal sphincters injury | 8 weeks
  Assessed by subsequent measures:
  1. Sphincter continuity in physical examination,
  2. Sphincter tension in physical examination,
  3. OASIS classification of perineal tears in transanal ultrasonography
  4. Starck scale for classification of anal sphincter injuries in transanal ultrasound (0-16 scale, no defect - 0; maximum - 16, means severe damage of both sphincters on a considerable length and circumference)
  5. Norderval scale for classification of anal sphincter injuries in transanal ultrasound (0-7 scale, no defect - 0, 7 is the maximal damage of both anal sphincters)
  6. anorectal manometry assessment to measure anal sphincters function
  All measurements are used to estimate the presence, extent and severity of anal sphincter injury.
  The main aim of the study is to establish whether the extension and severity of obstetric anal sphincter injury can be precisely assessed with parameters calculated from pelvic floor muscles using impedance spectroscopy.

SECONDARY OUTCOMES:
Adverse events | 8 weeks
  Evaluation of the frequency and intensity of adverse events associated with the use of the new diagnostic method.

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Surkont, MD, PhD, Principal Investigator — Centrum Medyczne Byc Kobieta s.c.
Locations (1):
- Centrum Medyczne Byc Kobieta s.c., Lodz, Łódź Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor's website — http://www.oasis-diagnostics.eu